CLINICAL TRIAL: NCT02313766
Title: Randomized Controlled Trial on Preoxygenation Through Spontaneous Breathing or Non Invasive Positive Pressure Ventilation With and Without Positive End Expiratory Pressure
Brief Title: Preoxygenation With Positive Inspiratory Pressure During Induction of Anesthesia
Acronym: PREOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2005-39
Record Dates: First submitted 2014-12-01; First posted 2014-12-10 (Estimated); Results first posted 2015-01-07 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Anesthesia
MeSH Terms: interventions — Intermittent Positive-Pressure Ventilation; Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- spontaneous breathing (SB) (No Intervention): preoxygenation through a face mask firmly applied and connected to the anaesthesia machine delivering a fresh gas flow of 12 l min-1. The inspired O2 concentration was set at 100%.
  End of preoxygenation FEO2=90%
- positive pressure ventilation (PPV) (Experimental): PPV : positive pressure ventilation : preoxygenation with noninvasive positive inspiratory pressure ventilation (12 cmH2O) without PEEP.
  Preoxygenation through a face mask firmly applied and connected to the anaesthesia machine - non invasive inspiratory ventilation mode - inspiratory trigger sensitivity was set at -2 l min-1, the adjustable pressure limiting valve was opened, and maximal airway pressure was limited at 18 cmH2O - PEEP=0 cmH2O End of preoxygenation FEO2=90%
  Interventions: Other: PPV : positive pressure ventilation
- PPV + PEEP (Experimental): PEEP : PPV + PEEP : preoxygenation with noninvasive positive inspiratory pressure ventilation (12 cmH2O) with PEEP at 6 cmH2O.
  Preoxygenation through a face mask firmly applied and connected to the anaesthesia machine - non invasive inspiratory ventilation mode - inspiratory trigger sensitivity was set at -2 l min-1, the adjustable pressure limiting valve was opened, and maximal airway pressure was limited at 18 cmH2O - PEEP=6 cmH2O End of preoxygenation FEO2=90%
  Interventions: Other: PEEP : PPV + PEEP

INTERVENTIONS:
Other: PPV : positive pressure ventilation — Inspiratory pressure support ventilation (12 cmH2O) without PEEP
  Arms: positive pressure ventilation (PPV)
Other: PEEP : PPV + PEEP — Inspiratory pressure support ventilation (12 cmH2O) with PEEP (6 cmH2O)
  Arms: PPV + PEEP

SUMMARY:
Adults patients scheduled for elective surgery were randomly allocated to receive preoxygenation with spontaneous breathing, positive pressure ventilation (positive inspiratory pressure: 12 cmH2O) without PEEP, and with PEEP (positive inspiratory pressure: 12 cmH2O, PEEP: 6 cmH2O). Preoxygenation time was measured from face mask positioning to FEO2=90% (FEO2 : expired fraction of O2). After endotracheal tube placement the time until SpO2=93% (SpO2 : peripheral oxygen saturation) was measured during monitored apnoea. Patient's discomfort was recorded (visual analogue scale).

DETAILED DESCRIPTION:
Inclusion criteria : age older 18 years, American Society of Anesthesiologists physical status I and II, and scheduled surgery with general anaesthesia and oro-tracheal intubation.

Exclusion criteria : rapid sequence induction, anticipated difficult mask ventilation (2 or more factors among age > 55 years, body mass index > 26 kg m-2, beard, history of snoring, lack of teeth), anticipated difficult intubation (history of difficult intubation, Mallampati class 3 and 4, thyromental distance < 60 mm, interincisor distance < 35 mm, limited cervical spine movement), and refusal to participate to the study and to sign informed consent.

Preoperative data recorded : age, height, weight, ASA physical status, and history of asthma, current smoking (ex-smokers were considered after a 3 month period without smoking), number of pack-years, sign inform consent The day of surgery, randomly allocation (random number table, block sizes of 15) to one of the 3 preoxygenation methods: spontaneous breathing, noninvasive positive inspiratory pressure ventilation (PPV) at 12 centimeters of water (cmH2O) without PEEP or with PEEP at 6 cmH2O (PEEP).

Intravenous line placement and standard monitoring. Preoxygenated through a face mask firmly applied and connected to the anaesthesia machine delivering a fresh gas flow of 12 l min-1. The circle breathing system was previously flushed with the O2 bypass during 30 s before mask placement. The inspired O2 concentration was set at 100%, the inspiratory trigger sensitivity was set at -2 l min-1, the adjustable pressure limiting valve was opened, and maximal airway pressure was limited at 18 cmH2O. Inspired and expired fraction of O2 and carbon dioxide (CO2) were continuously measured. End of the preoxygenation defined by FEO2=90%, intravenous anaesthesia was performed with propofol (2.5 mg kg-1 followed by a continuous administration at 8 mg kg-1 h-1 continuous infusion of propofol to target a bispectral index between 40 and 50), alfentanil 40 microg kg-1, and succinylcholine 1 mg kg-1. No face mask ventilation was provided before orotracheal intubation which was performed at the end of muscles fasciculation. The correct position of the tube (tracheal position above carina) was immediately checked using fiberoptic visualisation and was mandatory before atracurium 0.5 mg kg-1 administration. If tube misplacement occurred, the patient was excluded from the study in order to perform standard care. The time until SpO2 reached 93% was measured. The SpO2 and FEO2 were recorded every 10 s during the preoxygenation phase. The SpO2 was recorded every 10 s during the apnea phase.

Just before leaving the post-anaesthesia care unit, the patient was asked to evaluate the preoxygenation method with the following questions: How do you evaluate the preoxygenation phase on the scale (cursor placed on a 100 mm visual analogue scale) between very comfortable (0 mm) to very uncomfortable (100 mm)? Do you want to have the same preoxygenation method for further anaesthesia (yes/no)? Primary endpoint : time for preoxygenation (average 180 s) calculated from face mask positioning to FEO2=90%.

Secondary endpoints: duration of apnoea from tracheal tube positioning to SpO2 = 93% (average 5 to 10 min), and patient's comfort evaluated on a 0 to 100 mm visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I and II
* Scheduled surgery with general anaesthesia and oro-tracheal intubation

Exclusion Criteria:

* rapid sequence induction
* anticipated difficult mask ventilation
* anticipated difficult intubation
* refusal to participate to the study and to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual); Study Completion 2008-01 (Actual)

REFERENCES:
- [Derived] Hanouz JL, Lammens S, Tasle M, Lesage A, Gerard JL, Plaud B. Preoxygenation by spontaneous breathing or noninvasive positive pressure ventilation with and without positive end-expiratory pressure: A randomised controlled trial. Eur J Anaesthesiol. 2015 Dec;32(12):881-7. doi: 10.1097/EJA.0000000000000297. PMID 26225498

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned Recruitment period : from october 01,2006 to october 31,2007 The day of surgery, the patient was randomly allocated (random number table, equilibration block sizes of 15)
Pre-assignment Details: patients received oral information and signed a written informed consent at the end of the preanaesthesia medical consultation
Groups:
- Positive Pressure Ventilation (PPV): PPV : positive pressure ventilation : preoxygenation with noninvasive positive inspiratory pressure ventilation (12 cmH2O) without PEEP.
  Preoxygenation through a face mask firmly applied and connected to the anaesthesia machine - non invasive inspiratory ventilation mode - inspiratory trigger sensitivity was set at -2 l min-1, the adjustable pressure limiting valve was opened, and maximal airway pressure was limited at 18 cmH2O - PEEP=0 cmH2O End of preoxygenation FEO2=90%
  PPV : positive pressure ventilation: Inspiratory pressure support ventilation (12 cmH2O) without PEEP
- PPV + PEEP: PEEP : PPV + PEEP : preoxygenation with noninvasive positive inspiratory pressure ventilation (12 cmH2O) with PEEP at 6 cmH2O.
  Preoxygenation through a face mask firmly applied and connected to the anaesthesia machine - non invasive inspiratory ventilation mode - inspiratory trigger sensitivity was set at -2 l min-1, the adjustable pressure limiting valve was opened, and maximal airway pressure was limited at 18 cmH2O - PEEP=6 cmH2O End of preoxygenation FEO2=90%
  PEEP : PPV + PEEP: Inspiratory pressure support ventilation (12 cmH2O) with PEEP (6 cmH2O)
Period: Overall Study
Arm/Group | Spontaneous Breathing (SB) | Positive Pressure Ventilation (PPV) | PPV + PEEP
Started | 50 | 50 | 50
Completed | 49 | 47 | 50
Not Completed | 1 | 3 | 0
Not completed — surgery cancelled | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spontaneous Breathing (SB) | Positive Pressure Ventilation (PPV) | PPV + PEEP | Total
Number analyzed (Participants) | 49 | 47 | 50 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 42 | 42 | 41 | 125
  >=65 years | 7 | 5 | 9 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (18) | 40 (17) | 45 (20) | 44 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 20 | 66
  Male | 27 | 23 | 30 | 80
Region of Enrollment [Number; unit: participants]
  France | 49 | 47 | 50 | 146

OUTCOME MEASURES:

1. Primary Outcome: Time for Preoxygenationfrom Face Mask Positioning to FEO2=90%
Description: Time measured form face mask positioning until FEO2 reached 90% on the gas monitor
Time Frame: up to 5 min
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Spontaneous Breathing (SB) | Positive Pressure Ventilation (PPV) | PPV + PEEP
Number analyzed (Participants) | 49 | 47 | 50
seconds | 190 [130 to 264] | 153 [120 to 218] | 140 [100 to 200]

2. Secondary Outcome: Time Until SpO2=93%
Description: time until SpO2=93% after endotracheal tube placement has been confirmed
Time Frame: up to 10 min
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Spontaneous Breathing (SB) | Positive Pressure Ventilation (PPV) | PPV + PEEP
Number analyzed (Participants) | 49 | 47 | 50
seconds | 305 [263 to 383] | 370 [300 to 450] | 345 [245 to 435]

3. Secondary Outcome: Discomfort of the Preoxygenation Phase Self Reported by the Patient
Description: discomfort of the preoxygenation phase evaluated on a visual analogue scale (0 no discomfort - 100 maximal discomfort) just before PACU leaving
Time Frame: Before PACU leaving
Measure: Median (Inter-Quartile Range); unit: millimeters
Arm/Group | Spontaneous Breathing (SB) | Positive Pressure Ventilation (PPV) | PPV + PEEP
Number analyzed (Participants) | 49 | 47 | 50
millimeters | 0 [0 to 18] | 8 [0 to 20] | 0 [0 to 10]

ADVERSE EVENTS:
Arm/Group | Spontaneous Breathing (SB) | Positive Pressure Ventilation (PPV) | PPV + PEEP
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/47 | 0/50
Other Adverse Events (participants affected / at risk) | 1/49 | 0/47 | 0/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spontaneous Breathing (SB) (N=49) | Positive Pressure Ventilation (PPV) (N=47) | PPV + PEEP (N=50)
Anxiety (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Anxiety during face mask positioning for preoxygenation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes